CLINICAL TRIAL: NCT02347917
Title: A Phase I/II Clinical Study of BBI608 in Combination With Pemetrexed and Cisplatin in Adult Patients With Malignant Pleural Mesothelioma
Brief Title: A Study of BBI608 in Combination With Pemetrexed and Cisplatin in Adult Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8807005
Record Dates: First submitted 2015-01-21; First posted 2015-01-28 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Malignant Pleural Mesothelioma; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — napabucasin; Pemetrexed; Cisplatin

ARMS (1):
- BBI608 puls pemetrexed and cisplatin (Experimental)
  Interventions: Drug: BBI608; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: BBI608 — 480 mg orally twice daily (960 mg total daily dose)
Drug: Pemetrexed — 500 mg/m2 I.V. infusion on Day 1 of each treatment cycle (except for cycle 1, in which Pemetrexed will be given on Day 3).
Drug: Cisplatin — 75 mg/m2 I.V. infusion on Day 1 of each treatment cycle (except for Cycle 1, in which Cisplatin will be given on Day 3).

SUMMARY:
This is an open-label, multicenter, phase 1/2 study of BBI608 in combination with pemetrexed and cisplatin chemotherapy as a 1st line treatment for Malignant Pleural Mesothelioma (MPM).

ELIGIBILITY:
Phase 1

Inclusion Criteria:

* Histologically confirmed diagnosis of Malignant Pleural Mesothelioma (MPM) or Non-Small Cell Lung Cancer (NSCLC).
* Measurable disease as defined by the modified Response Evaluation Criteria in Solid Tumors (mRECIST) for MPM or the RECIST 1.1 for NSCLC.
* ≥ 20 years of age.
* Provision of written informed consent.
* For male or female patient of child producing potential: Must agree to use contraception or take measures to avoid pregnancy during the study and for 30 days after the last protocol treatment dose.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Hemoglobin (Hb) ≥ 9.0 g/dL.
* Neutrophils ≥ 1500/μL.
* Platelets ≥ 100,000/μL.
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5-fold the upper limit of normal range (ULN) [≤ 5-fold ULN with any liver metastasis].
* Total bilirubin ≤ 1.5-fold ULN.
* Creatinine clearance (estimated value) ≥ 60 mL/min.
* Life expectancy ≥ 3 months.
* Females of childbearing potential have a negative urine pregnancy test.

Phase 2

Inclusion Criteria:

* Histologically confirmed diagnosis of MPM.
* Treatment naïve and not indicated for resection.
* Measurable disease as defined by the modified RECIST.
* ≥ 20 years of age.
* Provision of written informed consent.
* For male or female patient of child producing potential: Must agree to use contraception or take measures to avoid pregnancy during the study and for 30 days after the last protocol treatment dose.
* ECOG Performance Status of 0 or 1.
* Hb ≥ 9.0 g/dL.
* Neutrophils ≥ 1500/μL.
* Platelets ≥ 100,000/μL.
* AST and ALT ≤ 2.5-fold ULN [≤ 5-fold ULN for patients with any liver metastasis].
* Total bilirubin ≤ 1.5-fold ULN.
* Creatinine clearance (estimated value) > 60 mL/min.
* Life expectancy ≥ 3 months.
* Females of childbearing potential have a negative urine pregnancy test.

Both Phase 1 and 2

Exclusion Criteria:

* Prior anti-cancer chemotherapy and radiotherapy.
* Prior hormonal therapy, immunotherapy, thermotherapy, operation.
* Any brain metastasis requiring treatment or symptomatic.
* Active multiple primary cancers.
* Crohn's disease, ulcerative colitis, small intestine resection.
* Abnormal ECGs.
* Prior myocardial infarction.
* Current use of antiarrhythmic medication.
* Uncontrolled concurrent diseases.
* Known severe hypersensitivity to pemetrexed, cisplatin or other drugs containing platinum.
* Women who are pregnant or breastfeeding.
* Received other investigational drugs.
* Unable or unwilling to swallow BBI608 capsules daily.
* Prior treatment with BBI608.
* Ineligible for participation in the study in the opinion of the Investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumitomo Pharma Co., Ltd. Japan, Study Director — Sumitomo Pharma Co., Ltd.
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Chiba
  - National Cancer Center Hospital, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study conducted from February 2015 to December 2017 and a total of 28 participants were enrolled at 9 medical institutions in Japan.
Pre-assignment Details: This clinical study consisted of two parts: Phase 1 and Phase 2. The study proceeded to Phase 2 part after Phase 1 part demonstrated the tolerability of BBI608 combined with Pem plus CDDP based on complete assessment of DLT. Participants were NOT enrolled in Phase 1 and Phase 2 in duplicate.
Groups:
- MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part); MPM: BBI608 + Pem + CDDP (Phase 2 Part): Participants orally received BBI608 (480 mg) twice daily plus intravenously received Pem (500 mg/m2) and CDDP (75 mg/m2) on Day 3 in only Cycles 1 and on Days 1 in Cycles 2 and subsequent cycles.
  Premeditation with folic acid and vitamin B12 was given to reduce occurrence of serious adverse drug reactions, with reference to the package insert for Pem. Each cycle was defined as 21 days.
Period: Overall Study
Arm/Group | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part)
Started | 4 | 24
Discontinued beforeBBI608 Administration | 0 | 0
Start BBI608 Administration | 4 | 24
Discontinued in DLT Evaluation Period (DLT was assessed in Phase 1 part only.) | 1 | 0
Complete DLT Evaluation Period (DLT was assessed in Phase 1 part only.) | 3 | 0
Discontinued After BBI608 Administration | 4 | 24
Discontinued Before Survival Observation | 0 | 1
Completed (Complete survival observation) | 4 | 23
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants were NOT enrolled in Phase 1 and Phase 2 in duplicate.
Groups:
- Total: Total of all reporting groups
Arm/Group | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) | Total
Number analyzed (Participants) | 4 | 24 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (5.00) | 65.6 (10.71) | 65.5 (9.854)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 22 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 24 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 24 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Primary cancer [Count of Participants; unit: Participants]
  MPM | 1 | 24 | 25
  NSCLC | 3 | 0 | 3
Weight [Mean (Standard Deviation); unit: kg] | 58.53 (10.278) | 63.11 (7.661) | 62.45 (8.025)
ECOG PS [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) performance status measures patients' disease status on the following scale: 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2=Ambulatory and capable of all selfcare, unable to carry out any work activities. Up and about >50% of waking hours; 3=Capable of only limited selfcare, confined to bed or chair >50% of waking hours; 4=Completely disabled. Totally confined to bed or chair; 5=Dead
  Participants
    0 | 3 | 11 | 14
    1 | 1 | 13 | 14
    2<= | 0 | 0 | 0
Disease classification [Count of Participants; unit: Participants] — Most types of cancer have four stages: stages I (1) to IV (4). Some cancers also have a stage 0 (zero). Lower stages indicate that the disease is more localized, or contained, whereas higher stages refer to cancers that have spread into other areas of the body: Stage 0 = cancer in situ, which means "in place"; Stage I = a small cancer or tumor that has not grown deeply into nearby tissues; Stage II and III = larger cancers or tumors that have grown more deeply into nearby tissue; Stage IV = the cancer has spread to other organs or parts of the body. Population: Of 4 participants in Phase 1 part, 3 participants with NSCLC and 1 participant with MPM enrolled.
  Participants
    MPM: number analyzed (Participants) | 1 | 24 | 25
    MPM: STAGE I | 0 | 0 | 0
    MPM: STAGE II | 0 | 2 | 2
    MPM: STAGE III | 0 | 5 | 5
    MPM: STAGE IV | 1 | 17 | 18
    NSCLC: number analyzed (Participants) | 3 | 0 | 3
    NSCLC: STAGE I | 0 | 0 | 0
    NSCLC: STAGE II | 0 | 0 | 0
    NSCLC: STAGE III | 0 | 0 | 0
    NSCLC: STAGE IV | 3 | 0 | 3
Tissue classification (MPM) [Count of Participants; unit: Participants] — Population: Of 4 participants in Phase 1 part, 3 participants with NSCLC and 1 participant with MPM enrolled.
  Participants
    number analyzed (Participants) | 1 | 24 | 25
    EPITHELIOID | 1 | 16 | 17
    SARCOMATOID | 0 | 3 | 3
    BIPHASIC | 0 | 5 | 5
    OTHER | 0 | 0 | 0
Tissue classification (NSCLC) [Count of Participants; unit: Participants] — Population: Of 4 participants in Phase 1 part, 3 participants with NSCLC and 1 participant with MPM enrolled.
  Participants
    number analyzed (Participants) | 3 | 0 | 3
    ADENOCARCINOMA | 3 | 0 | 3
    SQUAMOUS CELL CARCINOMA | 0 | 0 | 0
    LARGE CELL CARCINOMA | 0 | 0 | 0
    OTHER | 0 | 0 | 0
Metastases [Count of Participants; unit: Participants]
  Yes | 3 | 11 | 14
  No | 1 | 13 | 14
Disease duration [Mean (Standard Deviation); unit: month] | 3.91 (2.866) | 0.91 (0.726) | 1.34 (1.562)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Part: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Drug Reactions (ADRs)
Description: An AE is any untoward medical occurrence in a study subject administered an investigational drug and which does not necessarily have a causal relationship with this treatment.
  A SAE was an AE that met one or more of the following criteria:
  * Results in death
  * Is life-threatening
  * Requires hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability or incapacity
  * Is a congenital anomaly or birth defect
  * Is an important medical event that may jeopardize the subject or may require a medical or surgical intervention to prevent one of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization.
  An ADR was defined as adverse events assessed to be related to the investigational drug
Time Frame: Between initial dosing of the investigational drug and final evaluation in the follow-up observation period, about 17 months
Population: Safety analysis populations (Phase 1 part)
Measure: Count of Participants; unit: Participants
Arm/Group | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part)
Number analyzed (Participants) | 4
Participants
  Any AEs | 4
  AEs leading to death | 0
  Serious AEs | 0
  AEs leading to drug withdrawn (BBI608) | 1
  AEs leading to drug interrupted (BBI608) | 1
  AEs leading to dose reduced (BBI608) | 0
  Any ADRs | 4
  ADRs leading to death | 0
  Serious ADRs | 0
  ADRs leading to drug withdrawn (BBI608) | 1
  ADRs leading to drug interrupted (BBI608) | 1
  ADRs leading to dose reduced (BBI608) | 0

2. Primary Outcome: Phase 1 Part: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT was defined as an adverse event meeting any of the following that occurred during the DLT evaluation period in any participants given BBI608 with the causal relationship to BBI608 assessed as "Definite," "Probable," or "Possible." The severity of adverse events was graded according to the CTCAE v4.0-JCOG.
  * Grade 4 neutropenia persisting for ≥ 7 days
  * Grade ≥ 3 febrile neutropenia persisting for ≥ 5 days
  * Grade 3 thrombocytopenia requiring platelet transfusions, grade 4 thrombocytopenia
  * Grade ≥ 3 non-hematotoxicity except the following:
    1. Inappetence, nausea, vomiting and electrolyte abnormality which, within 3 days of onset, improved to grade ≤ 2 or resolved after appropriate treatment
    2. Diarrhoea and fatigue which, within 5 days of onset, improved to grade ≤ 2 or resolved after appropriate treatment
  * Other clinically significant signs in the opinion of the investigator
Time Frame: From Day 1 of Cycle 1 to Day 24 pre-dose examination (23 days)
Population: DLT evaluable population (3 participants with NSCLC in Phase 1 part)
  1 participant with MPM was excluded from DLT evaluable population because the BBI608 treatment compliance rate during DLT evaluation period did not meet the rate of 80% which of assessable for DLT and no adverse events assessed as DLT occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part)
Number analyzed (Participants) | 3
Participants | 0

3. Primary Outcome: Phase 1 Part: Maximum Observed Concentration (Cmax) and Minimum Observed Concentration (Cmin) of BBI608 When Administered With Pem and CDDP
Time Frame: Cycle 1 Day 1 (Cmax only) and Day 23
Population: Pharmacokinetic (PK) analysis population
  1 participant with MPM of 4 participants in the pharmacokinetic analysis population completed BBI608 administration on Day 14 in Cycle 1 and therefore was not included in the analysis for Cmax and AUC on Day 23.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part)
Number analyzed (Participants) | 4
ng/mL
  Day 1: Cmax | 307.5 [251 to 380]
  Day 23: Cmax: number analyzed (Participants) | 3
  Day 23: Cmax | 473.7 [316 to 643]
  Day 23: Cmin: number analyzed (Participants) | 3
  Day 23: Cmin | 196.1 [30.4 to 392.0]

4. Primary Outcome: Phase 1 Part: Area Under the Concentration-time Curve
Description: AUC0-12: Area under the concentration-time curve from time zero to 12 hours, AUC0-24: Area under the concentration-time curve from time zero to 24 hours, AUC0-inf: Area under the concentration-time curve from time zero to infinity
Time Frame: Cycle 1 Day 1 and Day 23
Population: as for outcome 3
Measure: Mean (Full Range); unit: h*ng/mL
Arm/Group | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part)
Number analyzed (Participants) | 4
h*ng/mL
  Day 1: AUC0-12 | 1814.3 [900 to 2443]
  Day 1: AUC0-24 | 2223.8 [1005 to 3060]
  Day 1: AUC0-inf | 2413.5 [1141 to 3536]
  Day 23: AUC0-12: number analyzed (Participants) | 3
  Day 23: AUC0-12 | 3797.0 [1788 to 5725]
  Day 23: AUC0-24: number analyzed (Participants) | 3
  Day 23: AUC0-24 | 6103.7 [1936 to 9948]
  Day 23: AUC0-inf: number analyzed (Participants) | 3
  Day 23: AUC0-inf | 10762.7 [1962 to 20834]

5. Primary Outcome: Phase 2 Part: Progression-free Survival (PFS)
Description: PFS was defined as the time from BBI608 administration to documented PD (as assessed according to the mRECIST or RECIST 1.1) or death, whichever is earlier. The result of imaging assessment by the imaging assessment committee was used for phase 2 part.
Time Frame: From BBI608 administration to documented PD or death, whichever is earlier, about 17 months
Population: modified ITT population. Efficacy was analyzed using the efficacy analysis population (i.e., modified ITT population; mITT), separately for Phase 1 part (n=4), Phase 2 part (n=24) and Phase 2 part including 1 participant with MPM in Phase 1 part (n=25).
Measure: Median (95% Confidence Interval); unit: month
Groups:
- MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part): Participants orally received BBI608(480 mg) twice daily plus intravenously received Pem (500 mg/m2) and CDDP (75 mg/m2) on Day 3 in only Cycles 1 and on Days1 in Cycles 2 and subsequent cycles.
  Premeditation with folic acid and vitamin B12 was given to reduce occurrence of serious adverse drug reactions, with reference to the package insert for Pem. Each cycle was defined as 21 days.
Arm/Group | MPM: BBI608 + Pem + CDDP (Phase 2 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part)
Number analyzed (Participants) | 24 | 25
month | 5.59 [2.89 to NA] — Not reached | 5.59 [2.89 to NA] — Not reached

6. Secondary Outcome: Best Overall Response
Description: The best overall response is the best response recorded from the start of the study treatment until the end of treatment. The RECIST 1.1 was used for the evaluation of tumor response and overall response in patients with NSCLC, and also the evaluation of any non-pleural lesions in patients with MPM. The mRECIST was used for the evaluation of tumor response and overall response in patients with MPM. The result of imaging assessment by study site was used for phase 1 part, and the result of imaging assessment by the imaging assessment committee was used for phase 2 part.
Time Frame: Every 6 weeks from the first dose of BBI608 until Week 30, and every 9 weeks from Week 31.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- NSCLC: BBI608 + Pem + CDDP (Phase 1 Part); MPM: BBI608 + Pem +CDDP (Phase 1 Part); MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part); MPM: BBI608 + Pem + CDDP (Phase 2 Part); MPM: BBI608 + Pem + CDDP (Phase 2 Part Including Participants With MPM in Phase 1 Part): Participants orally received BBI608 (480 mg) twice daily plus intravenously received Pem (500 mg/m2) and CDDP (75 mg/m2) on Day 3 in only Cycles 1 and on Days 1 in Cycles 2 and subsequent cycles.
  Premeditation with folic acid and vitamin B12 was given to reduce occurrence of serious adverse drug reactions, with reference to the package insert for Pem. Each cycle was defined as 21 days.
Arm/Group | NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem +CDDP (Phase 1 Part) | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including Participants With MPM in Phase 1 Part)
Number analyzed (Participants) | 3 | 1 | 4 | 24 | 25
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 0 | 8 | 8
  Stable disease (SD) | 3 | 0 | 3 | 11 | 11
  Progressive disease (PD) | 0 | 0 | 0 | 2 | 2
  Not evaluated (NE) | 0 | 1 | 1 | 3 | 4

7. Secondary Outcome: Response Rate (RR) and Disease Control Rate (DCR)
Description: Response rate (RR): Proportion of subjects whose best overall response is CR or PR.
  Disease control rate (DCR): Proportion of subjects whose best overall response is CR, PR or SD.
  The result of imaging assessment by study site was used for phase 1 part, and the result of imaging assessment by the imaging assessment committee was used for phase 2 part.
Time Frame: From BBI608 administration to death from any cause, about 17 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part): Participants orally received BBI608 (480 mg) twice daily plus intravenously received Pem (500 mg/m2) and CDDP (75 mg/m2) on Day 3 in only Cycles 1 and on Days 1 in Cycles 2 and subsequent cycles.
  Premeditation with folic acid and vitamin B12 was given to reduce occurrence of serious adverse drug reactions, with reference to the package insert for Pem. Each cycle was defined as 21 days.
Arm/Group | NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem +CDDP (Phase 1 Part) | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part)
Number analyzed (Participants) | 3 | 1 | 4 | 24 | 25
Participants
  Response rate (RR) | 0 | 0 | 0 | 8 | 8
  Disease control rate (DCR) | 3 | 0 | 3 | 19 | 19

8. Secondary Outcome: Overall Survival(OS)
Description: OS was defined as the time from BBI608 administration to death from any cause. Participants alive at final observation or lost to follow-up were censored at their last contact (i.e., visit or telephone) date.
Time Frame: From BBI608 administration to death from any cause, up to 31 months
Population: as for outcome 5
Measure: Median (Full Range); unit: month
Arm/Group | NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem +CDDP (Phase 1 Part) | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part)
Number analyzed (Participants) | 3 | 1 | 4 | 24 | 25
month | 19.81 [19.4 to 27.8] | 30.1 [30.1 to 30.1] | NA [19.4 to 30.1] — Not calculated for total population in Phase 1 part because calculated for each cancer type (i.e., NSCLC and MPM separately) | 12.14 [3.0 to 28.6] | 12.75 [3.0 to 30.1]

9. Secondary Outcome: Respiratory Function Tests (Vital Capacity [VC] and Forced Vital Capacity [FVC])
Time Frame: Every 6 weeks from the first dose of BBI608 until Week 30, and then every 9 weeks from Week 31 [Actually up to Week 111]
Population: modified ITT population. Efficacy was analyzed using the efficacy analysis population (i.e., modified ITT population; mITT), separately for Phase 1 part (n=4), Phase 2 part (n=24) and Phase 2 part including 1 participant with MPM in Phase 1 part (n=25). In respiratory function tests, data from 1 participant with MPM in Phase 1 part were not collected.
Measure: Median (Full Range); unit: mL
Arm/Group | NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem +CDDP (Phase 1 Part) | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part)
Number analyzed (Participants) | 3 | 0 | 4 | 24 | 25
mL
  The change from baseline in VC: 6 weeks: number analyzed (Participants) | 3 | 0 | 3 | 20 | 20
  The change from baseline in VC: 6 weeks | 70.0 [-10 to 200] |  | 70.0 [-10 to 200] | 30.0 [-470 to 410] | 30.0 [-470 to 410]
  The change from baseline in VC: 12 weeks: number analyzed (Participants) | 3 | 0 | 3 | 17 | 17
  The change from baseline in VC: 12 weeks | 110.0 [-90 to 140] |  | 110.0 [-90 to 140] | 0.0 [-370 to 940] | 0.0 [-370 to 940]
  The change from baseline in VC: 18 weeks: number analyzed (Participants) | 3 | 0 | 3 | 13 | 13
  The change from baseline in VC: 18 weeks | -60.0 [-70 to 90] |  | -60.0 [-70 to 90] | -70.0 [-700 to 1250] | -70.0 [-700 to 1250]
  The change from baseline in VC: 24 weeks: number analyzed (Participants) | 2 | 0 | 2 | 10 | 10
  The change from baseline in VC: 24 weeks | -290.0 [-630 to 50] |  | -290.0 [-630 to 50] | -50.0 [-570 to 1480] | -50.0 [-570 to 1480]
  The change from baseline in VC: 30 weeks: number analyzed (Participants) | 2 | 0 | 2 | 7 | 7
  The change from baseline in VC: 30 weeks | -240.0 [-510 to 30] |  | -240.0 [-510 to 30] | 20.0 [-530 to 1410] | 20.0 [-530 to 1410]
  The change from baseline in VC: 39 weeks: number analyzed (Participants) | 2 | 0 | 2 | 6 | 6
  The change from baseline in VC: 39 weeks | -305.0 [-600 to -10] |  | -305.0 [-600 to -10] | 30.0 [-660 to 870] | 30.0 [-660 to 870]
  The change from baseline in VC: 48 weeks: number analyzed (Participants) | 1 | 0 | 1 | 4 | 4
  The change from baseline in VC: 48 weeks | NA [-480 to -480] — because of 1 participant data only |  | NA [-480 to -480] — because of 1 participant data only | 15.0 [-100 to 910] | 15.0 [-100 to 910]
  The change from baseline in VC: 57 weeks: number analyzed (Participants) | 1 | 0 | 1 | 3 | 3
  The change from baseline in VC: 57 weeks | NA [-820 to -820] — because of 1 participant data only |  | NA [-820 to -820] — because of 1 participant data only | -20.0 [-70 to 1090] | -20.0 [-70 to 1090]
  The change from baseline in VC: 66 weeks: number analyzed (Participants) | 1 | 0 | 1 | 2 | 2
  The change from baseline in VC: 66 weeks | NA [-990 to -990] — because of 1 participant data only |  | NA [-990 to -990] — because of 1 participant data only | 300.0 [-110 to 710] | 300.0 [-110 to 710]
  The change from baseline in VC: 75 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in VC: 75 weeks |  |  |  | 175.0 [-400 to 750] | 175.0 [-400 to 750]
  The change from baseline in VC: 84 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in VC: 84 weeks |  |  |  | 145.0 [-580 to 870] | 145.0 [-580 to 870]
  The change from baseline in VC: 93 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in VC: 93 weeks |  |  |  | -205.0 [-890 to 480] | -205.0 [-890 to 480]
  The change from baseline in VC: 102 weeks: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  The change from baseline in VC: 102 weeks |  |  |  | NA [480 to 480] — because of 1 participant data only | NA [480 to 480] — because of 1 participant data only
  The change from baseline in VC: 111 weeks: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  The change from baseline in VC: 111 weeks |  |  |  | NA [280 to 280] — because of 1 participant data only | NA [280 to 280] — because of 1 participant data only
  The change from baseline in FVC: 6 weeks: number analyzed (Participants) | 3 | 0 | 3 | 20 | 20
  The change from baseline in FVC: 6 weeks | 0.0 [-50 to 120] |  | 0.0 [-50 to 120] | 35.0 [-380 to 390] | 35.0 [-380 to 390]
  The change from baseline in FVC: 12 weeks: number analyzed (Participants) | 3 | 0 | 3 | 17 | 17
  The change from baseline in FVC: 12 weeks | 80.0 [-110 to 90] |  | 80.0 [-110 to 90] | 10.0 [-400 to 1030] | 10.0 [-400 to 1030]
  The change from baseline in FVC: 18 weeks: number analyzed (Participants) | 3 | 0 | 3 | 13 | 13
  The change from baseline in FVC: 18 weeks | -20.0 [-110 to 0] |  | -20.0 [-110 to 0] | -140.0 [-860 to 1280] | -140.0 [-860 to 1280]
  The change from baseline in FVC: 24 weeks: number analyzed (Participants) | 2 | 0 | 2 | 10 | 10
  The change from baseline in FVC: 24 weeks | -155.0 [-390 to 80] |  | -155.0 [-390 to 80] | -50.0 [-610 to 1520] | -50.0 [-610 to 1520]
  The change from baseline in FVC: 30 weeks: number analyzed (Participants) | 2 | 0 | 2 | 7 | 7
  The change from baseline in FVC: 30 weeks | -265.0 [-570 to 40] |  | -265.0 [-570 to 40] | 150.0 [-430 to 1450] | 150.0 [-430 to 1450]
  The change from baseline in FVC: 39 weeks: number analyzed (Participants) | 2 | 0 | 2 | 6 | 6
  The change from baseline in FVC: 39 weeks | -345.0 [-530 to -160] |  | -345.0 [-530 to -160] | -35.0 [-530 to 770] | -35.0 [-530 to 770]
  The change from baseline in FVC: 48 weeks: number analyzed (Participants) | 1 | 0 | 1 | 4 | 4
  The change from baseline in FVC: 48 weeks | NA [-480 to -480] — because of 1 participant data only |  | NA [-480 to -480] — because of 1 participant data only | 70.0 [-160 to 800] | 70.0 [-160 to 800]
  The change from baseline in FVC: 57 weeks: number analyzed (Participants) | 1 | 0 | 1 | 3 | 3
  The change from baseline in FVC: 57 weeks | NA [-800 to -800] — because of 1 participant data only |  | NA [-800 to -800] — because of 1 participant data only | 60.0 [-70 to 880] | 60.0 [-70 to 880]
  The change from baseline in FVC: 66 weeks: number analyzed (Participants) | 1 | 0 | 1 | 2 | 2
  The change from baseline in FVC: 66 weeks | NA [-880 to -880] — because of 1 participant data only |  | NA [-880 to -880] — because of 1 participant data only | 300.0 [-140 to 740] | 300.0 [-140 to 740]
  The change from baseline in FVC: 75 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in FVC: 75 weeks |  |  |  | 50.0 [-550 to 650] | 50.0 [-550 to 650]
  The change from baseline in FVC: 84 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in FVC: 84 weeks |  |  |  | 10.0 [-580 to 600] | 10.0 [-580 to 600]
  The change from baseline in FVC: 93 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in FVC: 93 weeks |  |  |  | -230.0 [-900 to 440] | -230.0 [-900 to 440]
  The change from baseline in FVC: 102 weeks: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  The change from baseline in FVC: 102 weeks |  |  |  | NA [540 to 540] — because of 1 participant data only | NA [540 to 540] — because of 1 participant data only
  The change from baseline in FVC: 111 weeks: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  The change from baseline in FVC: 111 weeks |  |  |  | NA [490 to 490] — because of 1 participant data only | NA [490 to 490] — because of 1 participant data only

10. Secondary Outcome: Respiratory Function Tests (Forced Expiratory Volume in the First Second [FEV1])
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: L
Arm/Group | NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem +CDDP (Phase 1 Part) | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part)
Number analyzed (Participants) | 3 | 0 | 4 | 24 | 25
L
  The change from baseline in FEV1: 6 weeks: number analyzed (Participants) | 3 | 0 | 3 | 20 | 20
  The change from baseline in FEV1: 6 weeks | 0.160 [-0.01 to 0.16] |  | 0.160 [-0.01 to 0.16] | 0.050 [-0.40 to 0.33] | 0.050 [-0.40 to 0.33]
  The change from baseline in FEV1: 12 weeks: number analyzed (Participants) | 3 | 0 | 3 | 17 | 17
  The change from baseline in FEV1: 12 weeks | 0.070 [0.03 to 0.18] |  | 0.070 [0.03 to 0.18] | -0.130 [-0.33 to 0.52] | -0.130 [-0.33 to 0.52]
  The change from baseline in FEV1: 18 weeks: number analyzed (Participants) | 3 | 0 | 4 | 13 | 13
  The change from baseline in FEV1: 18 weeks | 0.000 [-0.13 to 0.16] |  | 0.000 [-0.13 to 0.16] | -0.110 [-0.56 to 0.63] | -0.110 [-0.56 to 0.63]
  The change from baseline in FEV1: 24 weeks: number analyzed (Participants) | 2 | 0 | 2 | 10 | 10
  The change from baseline in FEV1: 24 weeks | -0.010 [-0.16 to 0.14] |  | -0.010 [-0.16 to 0.14] | -0.040 [-0.45 to 0.78] | -0.040 [-0.45 to 0.78]
  The change from baseline in FEV1: 30 weeks: number analyzed (Participants) | 2 | 0 | 2 | 7 | 7
  The change from baseline in FEV1: 30 weeks | -0.055 [-0.23 to 0.12] |  | -0.055 [-0.23 to 0.12] | -0.030 [-0.29 to 0.71] | -0.030 [-0.29 to 0.71]
  The change from baseline in FEV1: 39 weeks: number analyzed (Participants) | 2 | 0 | 2 | 6 | 6
  The change from baseline in FEV1: 39 weeks | -0.140 [-0.28 to 0.00] |  | -0.140 [-0.28 to 0.00] | -0.050 [-0.37 to 0.26] | -0.050 [-0.37 to 0.26]
  The change from baseline in FEV1: 48 weeks: number analyzed (Participants) | 1 | 0 | 1 | 4 | 4
  The change from baseline in FEV1: 48 weeks | NA [-0.060 to -0.060] — because of 1 participant data only |  | NA [-0.060 to -0.060] — because of 1 participant data only | 0.115 [-0.12 to 0.39] | 0.115 [-0.12 to 0.39]
  The change from baseline in FEV1: 57 weeks: number analyzed (Participants) | 1 | 0 | 1 | 3 | 3
  The change from baseline in FEV1: 57 weeks | NA [-0.460 to -0.460] — because of 1 participant data only |  | NA [-0.460 to -0.460] — because of 1 participant data only | 0.010 [-0.07 to 0.31] | 0.010 [-0.07 to 0.31]
  The change from baseline in FEV1: 66 weeks: number analyzed (Participants) | 1 | 0 | 1 | 2 | 2
  The change from baseline in FEV1: 66 weeks | NA [-0.570 to -0.570] — because of 1 participant data only |  | NA [-0.570 to -0.570] — because of 1 participant data only | 0.085 [-0.16 to 0.33] | 0.085 [-0.16 to 0.33]
  The change from baseline in FEV1: 75 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in FEV1: 75 weeks |  |  |  | -0.045 [-0.42 to 0.33] | -0.045 [-0.42 to 0.33]
  The change from baseline in FEV1: 84 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in FEV1: 84 weeks |  |  |  | -0.130 [-0.44 to 0.18] | -0.130 [-0.44 to 0.18]
  The change from baseline in FEV1: 93 weeks: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2
  The change from baseline in FEV1: 93 weeks |  |  |  | -0.215 [-0.66 to 0.23] | -0.215 [-0.66 to 0.23]
  The change from baseline in FEV1: 102 weeks: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  The change from baseline in FEV1: 102 weeks |  |  |  | NA [0.150 to 0.150] — because of 1 participant data only | NA [0.150 to 0.150] — because of 1 participant data only
  The change from baseline in FEV1: 111 weeks: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  The change from baseline in FEV1: 111 weeks |  |  |  | NA [0.080 to 0.080] — because of 1 participant data only | NA [0.080 to 0.080] — because of 1 participant data only

ADVERSE EVENTS:
Time Frame: During a period from initial dosing of investigational drug to final evaluation in the follow-up observation period. up to 31 months for deaths, up to 11 months for Serious and Other (Not Including Serious) Adverse Events
Description: Safety analysis population [separately for Phase 1 part (n=4), Phase 2 part (n=24) and Phase 2 part including 1 participant with MPM in Phase 1 part (n=25)]
Arm/Group | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part)
All-Cause Mortality (participants affected / at risk) | 2/4 | 19/24 | 21/25
Serious Adverse Events (participants affected / at risk) | 0/4 | 7/24 | 7/25
Other Adverse Events (participants affected / at risk) | 4/4 | 24/24 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) (N=4) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) (N=24) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part) (N=25)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPM or NSCLC: BBI608 + Pem + CDDP (Phase 1 Part) (N=4) | MPM: BBI608 + Pem + CDDP (Phase 2 Part) (N=24) | MPM: BBI608 + Pem + CDDP (Phase 2 Part Including 1 Participant With MPM in Phase 1 Part) (N=25)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 14 (15) | 15 (16)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 14 (22) | 14 (22)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 24 (54) | 25 (55)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 5 (5) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (5) | 21 (49) | 22 (51)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 5 (5) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 12 (17) | 12 (17)
Face oedema (General disorders) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 2 (4) | 4 (10) | 4 (10)
Malaise (General disorders) | 1 (1) | 9 (11) | 9 (11)
Oedema peripheral (General disorders) | 0 (0) | 6 (11) | 6 (11)
Pyrexia (General disorders) | 0 (0) | 7 (9) | 7 (9)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 6 (6) | 6 (6)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 2 (3) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (7) | 12 (18) | 13 (19)
Platelet count decreased (Investigations) | 2 (6) | 4 (5) | 4 (5)
Weight decreased (Investigations) | 0 (0) | 6 (10) | 6 (10)
White blood cell count decreased (Investigations) | 2 (8) | 7 (11) | 8 (12)
Decreased appetite (Metabolism and nutrition disorders) | 3 (9) | 21 (45) | 22 (46)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 4 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 9 (13) | 9 (13)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (9) | 4 (9)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 6 (8) | 7 (9)
Headache (Nervous system disorders) | 1 (1) | 4 (10) | 4 (10)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (5) | 4 (5)
Chromaturia (Renal and urinary disorders) | 0 (0) | 4 (4) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 5 (6) | 5 (6)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 12 (22) | 13 (23)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT02347917/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT02347917/SAP_001.pdf